CLINICAL TRIAL: NCT01191346
Title: 3T Versus 1.5T MR Approaches in Target Definition for Malignant Gliomas: Is There a Significant Difference in Tumor Extent and Radiation Treatment Volume?
Brief Title: Radiation Planning Study for High Grade Brain Tumors
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Alison Kastl, BS, CCRC, Director of Clinical Trials, University of Cincinnati
Other Study IDs: BTC-G1
Record Dates: First submitted 2010-08-25; First posted 2010-08-30 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2014-12

CONDITIONS: High Grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3T MRI: Patients receiving 3T MRI
  Interventions: Other: 3T MRI

INTERVENTIONS:
Other: 3T MRI — 3T MRI in addition to standard 1.5T MRI for treatment planning

SUMMARY:
The purpose of this research study is to see if a higher strength MRI procedure provides better images to use in planning radiation treatments for patients with brain tumors in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed Grade III-IV glioma
* Planning to undergo radiation therapy

Exclusion Criteria:

* Grade I or II glioma
* Patients unable to undergo MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high grade glioma planning to receive radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Treatment volume | 1 year average
  To assess the difference in treatment volume for radiation planning in gliomas as calculated using 1.5T versus 3T magnets

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Guarnaschelli, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No